CLINICAL TRIAL: NCT04947020
Title: Multicenter Retrospective Trial for Analysis of Oncological Results of Patients with Primary Rectal Cancer Operated on Between 2013-2019
Brief Title: DataBase for Analysis of Rectal Cancer Oncological Results
Acronym: BARO
Status: Completed | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Radoslaw Pach, MD, PhD, Principal Investigator, Jagiellonian University
Other Study IDs: BARO Trial
Record Dates: First submitted 2021-06-24; First posted 2021-07-01 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Rectal Cancer; Metformin; Overall Survival; Lymph Node Metastases; Disease-free Survival
MeSH Terms: conditions — Rectal Neoplasms; Lymphatic Metastasis | interventions — Metformin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Rectal cancer: Patients with primary rectal cancer operated on between 2013 and 2019.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Metformin use before operation due to previously diagnosed diabetes.
  Other Names: Avamina; Etform; Formetic; Glucophage; Metfogamma; Metformax; Siofor; Symformin

SUMMARY:
The data will be obtained from 10 tertiary centers located in Poland (Cracow - coordinating center, Warsaw - 3 centers, Sosnowiec, Szczecin, Bydgoszcz, Lublin, Gdansk, Poznan) and 5 foreign centers.

The analyses will include patients with rectal cancer operated on between 2013-2019. A database in MS Excel is prepared that consists of following data:

* Type of neoadjuvant treatment (if any)
* Time-interval between the end of neoadjuvant treatment and surgery
* Type of surgery
* Staging of rectal cancer i.e. (y)pTNM
* Number of retrieved lymph nodes
* Number of lymph nodes with metastases
* R classification (R0, R1, R2)
* Preoperative medications (metformin, statins, NSAIDs, anticoagulants)
* Recurrence date and type (local, systemic, both diagnosed at the same time)
* Date of death or date of last follow-up visit

The aims of the study are following:

1. Establishing whether neoadjuvant treatment (PSCR or chemoradiotherapy) influences number of retrieved lymph nodes in rectal cancer
2. Establishing whether time-interval between the end of PSCR and surgery influences lymph node yield
3. Establishing the prognostic value of lymph node ratio - validation of the previously calculated cutoff point at the level of 0.41
4. Determining independent prognostic factors in rectal cancer - in particular related to medications taken before the operation, metformin and anti diabetic drugs in the first place

DETAILED DESCRIPTION:
Previously published studies showed that preoperative treatment of rectal cancer is associated with a lower number of lymph nodes retrieved during resection that is often lower than the recommended number of 12 nodes necessary for proper establishing of ypN category. A few studies revealed that lymph node ratio (LNR) is a more precise prognostic factor than pN category. The analysis conducted at the 1st Department of Surgery (Jagiellonian University, Cracow, Poland) based on patients' data from 1999 - 2006 year indicated that the median number of harvested lymph nodes after preoperative short course radiotherapy 5x5 Gy (PSCR) was 16. Therefore, PSCR did not seem to influence the number of lymph nodes in the operative specimen. Time-interval between radiotherapy and surgery (7-10 days versus 4-5 weeks) was not associated with lymph node yield, either.

Medication taken by the patients before operation may influence the treatment results as well. In a couple of studies metformin was identified as inhibitor of carcinogenesis according to antiangiogenic and antimetabolic effects and as a potential radiosensitizer. The anticancer property of metformin is largely attributed to its capability in modulating signaling pathways involved in cellular proliferation, apoptosis, and metabolism. In the last decade, mounting evidence supports the use of metformin in the prevention and treatment of colorectal cancer. Moreover, the use of metformin as monotherapy or as an adjuvant in colorectal cancer patients has led to further dose reduction and increased radio-chemosensitivity which lead to minimal gastrointestinal side effects and reduced toxicity. The use of metformin was associated with improved survival among colorectal cancer patients with type 2 diabetes mellitus compared to sulfonylureas and insulin. The effect of metformin in nondiabetic patients has not been evaluated so far. Based on the aforementioned results, it seems well-grounded to establish the influence of other medications (statins, nonsteroidal anti-inflammatory drugs, anticoagulants) on the results of combined treatment of rectal cancer with the assessment whether they are independent prognostic factors in comparison with such parameters as (y)pT, (y)pN or LNR.

After study initiation, a template of MS Excel database with manual will be sent to the Principal Investigators in every participating center. After obtaining the filled sheets from all participating centers, a central database will be prepared. No personal data of the patients (name, surname, personal ID numbers) will be collected and data in the central database will be anonymized.

Number of harvested lymph nodes will be compared in patients who underwent neoadjuvant chemoradiotherapy, PSCR, or surgery alone. In addition, number of retrieved lymph nodes and lymph node ratio will be compared in patients operated on after different time-intervals between PSCR and surgery (< 7 days and > 4 weeks). Kaplan-Meier curves will be drawn to established influence of number and ratio of harvested lymph nodes on overall survival and disease-free survival. Local and systemic recurrence rate will be established and compared in analysed patients. Statistical analysis will be performed with SPSS 27 for Mac. Variables without normal distribution will be compared by means of Mann Whitney U and Chi-square tests. Cumulative proportions of surviving will be compared with the use of log-rank test. Univariate and multivariate Cox regression will be performed to establish prognostic factors in analysed population.

The study is academic and non-commercial. The participating centers will not have to cover any additional cost as the treatment options analysed constitute standard clinical practice. No financial support is granted for investigators nor study participants.

ELIGIBILITY:
Inclusion Criteria:

* Primary rectal cancer confirmed histologically
* Age ≥ 18

Exclusion Criteria:

* Recurrent rectal cancer
* Oncological radicalization after previous local excision of rectal cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with primary rectal cancer operated on between 2013 and 2019.
Sampling Method: Non-Probability Sample
Enrollment: 2443 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Overall survival | 3 years
  Overall survival of analysed patients

SECONDARY OUTCOMES:
Disease-free survival | 3 years
  Disease-free survival of analysed patients

OTHER OUTCOMES:
Lymph node yield | 3 years
  Lymph node yield in analysed patients
Lymph node ratio | 3 years
  Metastatic to all retrieved lymph node ratio

CONTACTS AND LOCATIONS:
Overall Officials: Radoslaw Pach, PhD, Principal Investigator — Jagiellonian University; Antoni Szczepanik, PhD, Study Chair — Jagiellonian University
Locations (1):
- 1st Department of General Surgery, Krakow, Malopolska, Poland

IPD SHARING:
Plan to Share IPD: No
Anonimized database will be shared only with researchers participating in the study.